CLINICAL TRIAL: NCT00659633
Title: The Effect of Intravenous Lidocaine on Allodynia (Carl Koller Grant)
Brief Title: The Effect of Intravenous Lidocaine on Allodynia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Society of Regional Anesthesia (Other)
Responsible Party: Principal Investigator, Michael Froelich, Associate Proffesor Anesthesiology M.D., University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F061204014
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-06

CONDITIONS: Pain
Keywords: lidocaine; allodynia; chronic regional pain syndrome; pain
MeSH Terms: conditions — Pain; Hyperalgesia; Complex Regional Pain Syndromes | interventions — Lidocaine; Lidoderm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lidocaine (Experimental): Intravenous lidocaine for neuropathic pain
  Interventions: Drug: lidocaine

INTERVENTIONS:
Drug: lidocaine — intravenous, effect site concentration: 2mcg/ml, 15-20 min infusion, once
  Other Names: Lidoderm; Xylocaine

SUMMARY:
The purpose of this study is to study if lidocaine, given intravenously, reduces pain.

DETAILED DESCRIPTION:
Clinicians use lidocaine intravenously in a fashion that suggests that it might have analgesic effects. Therefore, we test the hypothesis that lidocaine reduces pain intensity in response to experimental pain.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Regional Pain Syndrome diagnostic criteria by the Work Safe BC. vi

Exclusion Criteria:

* History of Substance abuse
* Other Medications: CRPS patients are expected to be treated for chronic pain, whether the current treatment regimen interferes with sensory motor testing will be determined on a case by case basis.
* Coronary Artery Disease (CAD): unstable
* Congestive Heart Failure (CHF): unstable
* Heart Arrhythmia: symptomatic
* Chronic Obstructive Pulmonary Disease (COPD)
* Lidocaine Allergy
* Diagnostic and Statistical Manual of Mental Disorders (Rev IV): Axis I: Common Axis I disorders include depression, anxiety disorders, bipolar disorder, ADHD, and schizophrenia. Axis II: borderline personality disorder, schizotypal personality disorder, antisocial personality disorder, and mild mental retardation.
* Presence of Contraindications for MRI
* Presence of electronically, magnetically, and mechanically activated implants
* Electronically, magnetically, and mechanically activated implants
* Ferromagnetic or electronically operated active devices like automatic cardioverter defibrillators
* Cardiac pacemakers
* Metallic splinters in the eye
* Ferromagnetic haemostatic clips in the central nervous system (CNS)
* Claustrophobia
* Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-12; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Froelich, MD, MS, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lidocaine
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lidocaine
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Pain Perception
Description: Assessing heat pain perception (pain intensity) before, during, and after lidocaine infusion by means of patient self-report using a mechanical slide algometer.
  The mechanical slide algometer [Price et al. (1994)] looks like a ruler that exposes a red bar with the end-points: no pain (left) and most pain imaginable (right). The use the slider to express their perceived pain. On the back of the ruler a numerical scale ranging from 0 (no pain) to 10 (worst imaginable pain) translates the patient's rating into a numeric scale.
Time Frame: Participants will be followed from baseline through 128 minutes
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lidocaine
Number analyzed (Participants) | 10
units on a scale
  Baseline | 5.40303 (0.72232)
  Infusion | 5.1457 (0.72050)
  After Infusion | 5.13171 (0.72141)

ADVERSE EVENTS:
Arm/Group | Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No